CLINICAL TRIAL: NCT00545506
Title: The Influence of a Warmed Surgical Bandage System on Subcutaneous Tiisue Oxygen Tension After Cardiac Surgery
Brief Title: The Influence of a Warmed Surgical Bandage System on Subcutaneous Tissue Oxygen Tension After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of eligible patients
Sponsor: Medical University of Vienna (Other)
Collaborators: Outcomes Research Consortium (Other)
Responsible Party: Principal Investigator, Helmut Hager, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1.0
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Surgery
Keywords: wound infection; tissue oxygen tension; local warming
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional bandage (Active Comparator): conventional bandage on sternal wound after skin closure after cardiac surgery. conventional gauze covered with elastic adhesive (Medipore™ Dress-it) The designated bandage will be positioned in the operating room by the surgeons after the skin will be closed. The conventional elastic bandage consists of several layers of gauze covered with a special adhesive bandage
  Interventions: Device: conventional bandage
- warming bandage (Active Comparator): The Warm-Up bandage consists of an adhesive shell and a foam frame that supports a clear window about one cm above the surface of the wound. A battery-powered heating card can then be inserted into the window to provide gentle warming of the wound. The surface temperature of heating card is fixed at 38°C, and heat is usually provided for two hours at a time. That is, the experimental bandage will be continuously applied to the wound and heated to 38°C using a two-hour on/off cycle.
  Interventions: Device: warming bandage

INTERVENTIONS:
Device: conventional bandage
  Arms: conventional bandage
Device: warming bandage
  Arms: warming bandage

SUMMARY:
Warmed Surgical Bandage may improve tissue oxygenation and thus on the long run reduce wound infections

DETAILED DESCRIPTION:
Wound infections are common and serious complications of anesthesia and surgery. The morbidity associated with surgical infections is considerable and includes substantial prolongation of hospitalization.

The wound infection risk in patients undergoing cardiac surgery ranges from 0.8 to 17.7% including both superficial and deep sternal infections.

Major factors influencing the incidence of surgical wound infection other than site and complexity of surgery, underlying illness, timely administration of prophylactic antibiotics, intraoperative patient temperature, hypovolemia and tissue oxygen tension. The primary determinant of tissue oxygen availability is local perfusion. Thermoregulatory status is one of the major factors influencing tissue perfusion. Local warming induces pre- capillary vasodilation and improves tissue oxygenation. Local warming of surgical wounds may provide a simple and inexpensive way to reduce perioperative wound complications. Specifically, we will test the hypothesis that Warm- Up therapy increases postoperative tissue oxygen tension in patients undergoing cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age scheduled for elective cardiac surgery on normothermic cardio-pulmonary bypass will be invited to participate

Exclusion Criteria:

* Emergency surgery
* Pre - or postoperative on intraaortic balloon pump
* Preoperative mechanical ventilation
* Postoperative respiratory failure
* Postoperative extracorporal membrane oxygenation
* Left ventricular function < 40%
* Fever (core temperature > 38 °C) or current infection
* No anticipated or no definitive primary closure of surgical wound.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Kabon, MD, Principal Investigator — Medical University Vienna,Spitalgasse 23, 1090 Vienna, Austria; Helmut Hager, MD, Principal Investigator — Medical University Vienna, Spitalgasse 23, 1090 Vienna, Austra
Locations (1):
- Medical University Vienna, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: research personnel will screen the patient list one day before surgery to identify eligible patients
Groups:
- Heart Surgery, Wound Infection, Conventional Bandage: konventional bandage (conventional gauze covered with elastic adhesive (Medipore™ Dress-it)) on sternal wound
- Heart Surgery, Wound Infection, Warming Bandage, Tissue Oxygen: warming bandage on sternal wound The Warm-Up bandage consists of an adhesive shell and a foam frame that supports a clear window about one cm above the surface of the wound. A battery-powered heating card can then be inserted into the window to provide gentle warming of the wound. The experimental bandage will be continuously applied to the wound and heated to 38°C using a two-hour on/off cycle
Period: Overall Study
Arm/Group | Heart Surgery, Wound Infection, Conventional Bandage | Heart Surgery, Wound Infection, Warming Bandage, Tissue Oxygen
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heart Surgery, Wound Infection, Conventional Bandage | Heart Surgery, Wound Infection, Warming Bandage, Tissue Oxygen | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (5) | 55 (5) | 55 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  Austria | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Tissue Oxygen Tension in the Sternal Wound
Description: Tissue oxygen tension in the wound Tissue oxygen tension will be measured with a polarographic electrode system (Licox CMP, GMS Germany), the oxygen electrode will be calibrated with room air (154 mmHg) and then positioned within the silastic tonometer that will be inserted 2 3 cm lateral to the surgical incision.
Time Frame: 8 hours
Population: It was not possible to analyse the data because there was not enough data from the recruited population.
Arm/Group | Heart Surgery, Wound Infection, Conventional Bandage | Heart Surgery, Wound Infection, Warming Bandage, Tissue Oxygen
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Heart Surgery, Wound Infection, Conventional Bandage | Heart Surgery, Wound Infection, Warming Bandage, Tissue Oxygen
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
Tissue oxygen tension maybe difficult to measure in the sternal wound

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes